CLINICAL TRIAL: NCT04332419
Title: Comparison of Yttrium-90 Absorbed Doses Using PET/CT Versus PET/MR Imaging in Patients Undergoing Selective Internal Radiation Therapy for Hepatic Malignancies
Brief Title: Comparison of Yttrium-90 Absorbed Doses Using PET/CT Versus PET/MR Imaging for Hepatic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE13219
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Hepatic Malignancies
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography; Sirtuins; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PET/CT & PET/MR (Experimental): One-time PET/MR imaging in addition to the standard PET/CT imaging, both performed on the same day of the treatment procedure (Selective Internal Radiation Therapy Y-90 RE). Participants will be randomized to receive either of the imaging modalities first, based on the availability of the imaging device, and less than 1 hour apart.
  Interventions: Device: PET/CT; Device: PET/MR; Radiation: SIRT with Y-90

INTERVENTIONS:
Device: PET/CT — Standard Imaging
Device: PET/MR — Additional Imaging
Radiation: SIRT with Y-90 — SIRT with Y-90 for palliative treatment of the liver malignancy.

SUMMARY:
The purpose of this study is to compare the results of positron emission tomography/computer tomography (PET/CT) to positron emission tomography/magnetic resonance imaging (PET/MRI) to help determine any added advantage of one over the other in relation to a tumor which might assist in further management plans.

DETAILED DESCRIPTION:
Participants in this study will undergo PET/CT (standard imaging) and PET/MR (additional imaging), within 6 hours after SIRT with Y-90 for palliative treatment of the liver malignancy. Patients will be randomized to receive either of the imaging modalities first, based on the availability of the imaging device, and less than 1 hour apart. Upon acquirement and construction of PET/CT and PET/MR images, a software (MIM SurePlan LiverY90) would be utilized for semi-automatic determination of the liver/tumor contours and calculation of the Y-90 absorbed doses (Gy) in the regions of interest (including within tumor and background liver outlines) using the Local Deposition Method.

The primary objective of this study is to assess the agreement between post-Y-90 RE absorbed doses (Gy) in the liver tumor tissues based on PET/CT versus PET/MR imaging. This would permit the comparison of Y-90 tumor absorbed doses, acquired from PET/MR, with the current standard of care PET/CT imaging to verify the data consistency and to validate its application for the prediction of tumor response to treatment.

The secondary objective of this study is to assess the agreement between post-Y-90 RE absorbed doses (Gy) in the background liver tissues (surrounding tumors), based on PET/CT versus PET/MR imaging. This would permit the comparison of Y-90 background liver absorbed doses, acquired from PET/MR, with the current standard of care PET/CT imaging to verify the data consistency and to validate its application for the prediction of dose toxicity.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a liver malignancy and is scheduled for SIRT with Y-90; AND
* The patient is an adult, self-competent, and able to provide informed consent to participate in the study

Exclusion Criteria:

* The patient loses competence, has a condition that questions their ability to provide informed consent independently (e.g. cannot communicate in English), or withdraws consent to participate within any time in the study period; OR
* The patient is not eligible to undergo MRI due to the presence of metal devices or implants in their body; OR
* Both imaging modalities cannot take place within 6 hours after Y-90 RE; OR
* Both imaging modalities cannot take place within 1 hour apart from each other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ram Gurajala, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Team will be sharing study results but not IPD because of HIPAA regulations

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET/CT & PET/MR
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | PET/CT & PET/MR
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Reproducibility Coefficient (RDC) Between the Two Imaging Modalities in Liver Tumor Tissues
Description: RDC between the two imaging modalities for post-Y-90 Radioembolization (RE) absorbed doses (Gy) in the liver tumor tissues The RDC is the minimum difference between the two measurements that can be considered a true difference, with 95% confidence.
Time Frame: Post-op day 0, 1 hour apart
Measure: Mean (95% Confidence Interval); unit: percent difference
Units Other Than Participants: Tumors
Arm/Group | PET/CT & PET/MR
Number analyzed (Participants) | 11
Number analyzed (Tumors) | 17
percent difference | 16.9 [12.7 to 25.3]

2. Secondary Outcome: RDC Between the Two Imaging Modalities in Background Liver Tissues
Description: RDC between the two imaging modalities for post-Y-90 RE absorbed doses (Gy) in the background liver tissues
  The RDC is the minimum difference between the two measurements that can be considered a true difference, with 95% confidence.
Time Frame: Post-op day 0, 1 hour apart
Measure: Mean (95% Confidence Interval); unit: percent difference
Units Other Than Participants: sessions
Arm/Group | PET/CT & PET/MR
Number analyzed (Participants) | 11
Number analyzed (sessions) | 17
percent difference | 25.8 [18.5 to 42.5]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | PET/CT & PET/MR
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT04332419/Prot_SAP_002.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04332419/ICF_001.pdf